CLINICAL TRIAL: NCT03322839
Title: Implementing the Swedish Guideline for the Prevention of Common Mental Disorders at the Workplace in Schools: Study Protocol of a Cluster Randomized Controlled Trial Using Multifaceted Implementation Strategies
Brief Title: Evaluating the Effectiveness of Multifaceted Implementation Strategies for Implementing a Guideline for the Prevention of Common Mental Disorders at the Workplace in Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lydia Kwak, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150571; 150571 (Other Grant/Funding Number: AFA-insurance)
Record Dates: First submitted 2017-09-19; First posted 2017-10-26 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Common Mental Disorders
Keywords: Guideline-adherence; Implementation; Implementation-strategies; Randomized-controlled-trial; Organisational risk-factors; Schools; Social risk-factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifaceted implementation strategies (Experimental): The school-management will participate in a one-day training. In addition each intervention school will form an implementation team that is responsible for the implementation of the guideline within their school. The implementation teams will participate in 4-5 workshops in order to support the implementation process.
  Interventions: Behavioral: Multifaceted implementation strategies
- Single implementation strategy (Active Comparator): The control-schools will only receive training to the school-management.
  Interventions: Behavioral: Single implementation strategy

INTERVENTIONS:
Behavioral: Multifaceted implementation strategies — The school-management will participate in a one-day training aimed at providing knowledge and skills related the recommendations of the guideline for the prevention of common mental disorders at the workplace.In addition every intervention school will form an implementation team that is responsible for the implementation of the guideline. The implementation team will comprise of approximately 3-5 individuals with experience in the field of social and organizational work environment, for example school-management and occupational health and safety representative. The implementation teams will participate in 4-5 workshops aimed at supporting the implementation process. Intervention schools within the same municipality will participate in the same workshop in order to promote peer-support.
  Arms: Multifaceted implementation strategies
Behavioral: Single implementation strategy — The school-management will participate in a one-day training aimed at providing knowledge and skills related to the recommendations of the guideline for the prevention of common mental disorders at the workplace
  Arms: Single implementation strategy

SUMMARY:
Given today's high prevalence of common mental disorders and related sick leave among teachers an urgent need exists for a more sustainable working life for this professional group. One way of doing this is by improving schools' social and organizational risk management. Recent reports have shown that many schools in Sweden however lack a structured approach to the management of social and organizational risks. In 2015, we launched the first Swedish occupational health guideline to support a structured prevention of social and organizational risks at the workplace with the aim of preventing common mental disorders. The long-term goal of this study is to support the implementation of this guideline within schools in order to improve social and organizational risk management and in doing so reduce risk factors for mental ill-health and related sick days. The objective of the study is to fill the current research-to-practice gap by conducting a cluster-randomized controlled trial that compares the effectiveness of two implementation strategies for implementing the guideline in schools. The strategies that will be compared are training (ARM 1) versus training in combination with implementation teams and workshops (ARM 2). Our hypothesis for the study is that schools that receive support in implementing the guideline through combined strategies are more responsive to working in a structured and systematic manner with the management of social and organizational risks than schools that only receive training. The trial will be conducted in 20 primary schools in two municipalities in Sweden. All schools have agreed to participate. The primary outcomes are adherence to the guideline (implementation effectiveness) and self-reported exhaustion among schools personnel (intervention effectiveness); the secondary outcomes are risk factors for mental ill-health and absenteeism. Data will be collected at baseline, 6, 12 and 24 months by mixed methods (i.e. survey, focus-group interviews, observation, and register-data).

ELIGIBILITY:
Inclusion Criteria:

* all individuals who are employed by the participating schools

Exclusion Criteria:

* individuals employed by the participating municipalities and not by the participating schools, for example cleaning personal. Individuals on sick-leave

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Guideline adherence (implementation effectiveness) | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in adherence to the recommendations of the guideline during 6, 12 and 24 months follow-up period. We will use a questionnaire directed at the school management and a questionnaire directed at the school personnel. The questionnaires contain statements related to the recommendations in the guideline, such as "at our school we have clear and practical policies for preventing mental ill-health among our employees".
Exhaustion (intervention effectiveness) | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in personnel's self-reported exhaustion during 6, 12 and 24 months follow. We hypothesize that adherence to the recommendations of the guideline will affect school personnel's self-reported exhaustion assessed with the Oldenburg Burnout Inventory (response format 1-4).

SECONDARY OUTCOMES:
Psychosocial safety climate | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported psychosocial safety climate as assessed by the 11-items of the Psychosocial Safety Climate Scale (response format 1-5)
Job demands | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported job-demands as assessed by 11 items of the Copenhagen Psychosocial Questionnaire (response form 1-5)
Influence at work | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported influence at work as assessed by 4 items of the Copenhagen Psychosocial Questionnaire (response-form 1-5)
Social support colleagues | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported social support as assessed by 3 items of the Copenhagen Psychosocial Questionnaire (response-form 1-5)
Possibilities for development | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported possibilities for development as assessed by 4 items of the Copenhagen Psychosocial Questionnaire (response-form 1-5)
Commitment to the workplace | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported commitment as assessed by 3 items of the Copenhagen Psychosocial Questionnaire (response-form 1-5)
Social support superior | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported social support from superior as assessed by 3 items of the Copenhagen Psychosocial Questionnaire (response-form 1-5)
Work engagement | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported engagement as assessed by 3 items of the Utrecht Work Engagement Scale (response-form 1-7)
Self-perceived health | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-perceived health as assessed with a single question (response-form 1-5)
Self-reported stress | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported stress as assessed with a single question (response-form 1-5)
Work-family conflict | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported work-family conflict as assessed with 4 items of the Copenhagen Psychosocial Questionnaire (response-form 1-4)
Recovery | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported recovery as assessed with 1 item (response-form 1-5)
Work performance impairment due to health problems | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in work performance as assessed by a question based on one item from the Work productivity Activity impairment - General Health Questionnaire (response format 0-10)
Work performance impairment due to problems in the work environment | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in work performance as assessed by a question based on one item from the Work Productivity Activity Impairment - General Health Questionnaire (response format from 0-10)
Self-reported sickness absenteeism | At baseline and 6, 12 and 24 months after baseline
  Change from baseline in self-reported sickness absenteeism as assessed by 2 items
Registered sickness absenteeism | 12 months prior to baseline, and during 24 months after baseline
  Change in total sick-leave due to common mental disorders in days, register data (sickness benefit and disability pension).
Recognition (reward) | At baseline and 6, 12 and 24 months after baseline
  Change from baseline self-reported collaboration and leadership as assessed by 3-items of Copenhagen Psychosocial Questionnaire (response-format 1-5)
Self-reported stress (SMS) | Measured every 4th week over 12 months from baseline
  Change from baseline in self-reported stress as assessed by one item sent by text-message by mobile-phone
Process evaluation data | Assessed during the 24 month study period.
  Process data will be collected over the 24 months. This data will be assessed by focus-group interviews.
Process evaluation data | Assessed during the 24 month study period.
  Process data will be collected over the 24 months. This data will be assessed by questionnaires
Process evaluation data | Assessed during the 24 month study period.
  Process data will be collected over the 24 months. This data will be assessed by observation
Process evaluation data | Assessed during the 24 month study period.
  Process data will be collected over the 24 months. This data will be assessed by documentation.
Barriers | Assessed during the 24 month study period
  Information will be collected on possible barriers that may have influenced the implementation process. This data will be assessed by focus-group interviews
Barriers | Assessed during the 24 month study period
  Information will be collected on possible barriers that may have influenced the implementation process. This data will be assessed by questionnaires
Barriers | Assessed during the 24 month study period
  Information will be collected on possible barriers that may have influenced the implementation process. This data will be assessed by observation
Barriers | Assessed during the 24 month study period
  Information will be collected on possible barriers that may have influenced the implementation process. This data will be assessed by documentation.
Facilitators | Assessed during the 24 month study period
  Information will be collected on possible facilitators that may have influenced the implementation process. This data will be assessed by focus-group interviews
Facilitators | Assessed during the 24 month study period
  Information will be collected on possible facilitators that may have influenced the implementation process. This data will be assessed by questionnaires
Facilitators | Assessed during the 24 month study period
  Information will be collected on possible facilitators that may have influenced the implementation process. This data will be assessed by observation
Facilitators | Assessed during the 24 month study period
  Information will be collected on possible facilitators that may have influenced the implementation process. This data will be assessed by documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Kwak, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Unit for Intervention and Implementation Research for Worker Health, Institute for Environmental Medicine, Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The ethical approval does not allow data-sharing of individual participation data.

REFERENCES:
- [Derived] Kwak L, Lornudd C, Bjorklund C, Bergstrom G, Nybergh L, Elinder LS, Stigmar K, Wahlin C, Jensen I. Implementation of the Swedish Guideline for Prevention of Mental ill-health at the Workplace: study protocol of a cluster randomized controlled trial, using multifaceted implementation strategies in schools. BMC Public Health. 2019 Dec 11;19(1):1668. doi: 10.1186/s12889-019-7976-6. PMID 31829186